CLINICAL TRIAL: NCT04838717
Title: A Randomized Non-Inferiority Clinical Trial of Doxycyline Vs BPG for Early Syphilis
Brief Title: Clinical Trial of Doxycycline VS BPG for Early Syphilis (SY-DOXY)
Acronym: SY-DOXY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180588; 2019-003278-21 (EudraCT Number)
Record Dates: First submitted 2021-01-29; First posted 2021-04-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Syphilis
Keywords: early syphilis; Doxycycline; Benzathine benzyl penicillin G
MeSH Terms: conditions — Syphilis | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BPG Arm (Active Comparator): BPG injections will be performed at the participating center
  Interventions: Drug: BPG; Drug: Doxycycline
- Doxycycline Arm (Experimental): Dispensing of Doxycycline 100 mg is carried out at one time at V0 - Inclusion visit.
  Interventions: Drug: BPG; Drug: Doxycycline

INTERVENTIONS:
Drug: BPG — intramuscular injection of 2.4 million units
Drug: Doxycycline — Oral: at a dose of 100 mg bid for 14 days

SUMMARY:
According to European and US Centers for Disease Control and Prevention (CDC) guidelines, the recommended treatment for uncomplicated early syphilis in adults (i.e. primary, secondary and early latent) is a single intramuscular injection of 2.4 million units of benzathine benzylpenicillin G (BPG). Recent reviews have also recommended BPG as the first-line treatment of early syphilis, reporting a success rate of more than 90% over a large panel of studies. This form of the drug provides weeks of treponemicidal levels of penicillin in the blood, but does not efficiently cross the blood-brain barrier.

However, despite the use of BPG for almost 70 years and its status as the gold standard treatment for early syphilis, the need to administer this antibiotic parenterally has led to the use of second-line oral antibiotics, including firstgeneration macrolides, and then second-generation macrolides, such as azithromycin. Several African studies have shown 1 g azithromycin bid treatment for one day to be effective against early syphilis, but most authors agree that azithromycin should not generally be used as resistance to this macrolide is highly prevalent in Western countries. Moreover, a recent study by our group showed that more than 80% of the treponemal strains isolated in France harbor the mutation conferring resistance to azithromycin. The use of this alternative would, therefore, be highly unlikely to be effective in France. Tetracycline antibiotics have also been proposed as an alternative in patients with a contraindication for BPG or other forms of penicillin. Doxycycline, at a dose of 100 mg orally twice daily for 14 days, has been endorsed as a preferred alternative treatment, but few data are available concerning its efficacy. This issue is crucial, for two main reasons: there has been a recrudescence of early syphilis in most western countries over the last 20 years, increasing the need for BPG, and two periods of BPG shortage were experienced in 2013 and 2017, leading to the use of alternative treatments due to the temporary unavailability of BPG or its limitation to cases in which no other treatment was possible. Data for the manufacturing and distribution of antibiotics are not publicly available, but reports of limited availability, shortages, and price increases for old antibiotics suggest that the current system is too fragile to provide what should be a given in modern medicine: access to effective treatment for common and potentially severe bacterial infections. The recurrence of BPG shortages over the last five years has created an urgent need to demonstrate that doxycycline is safe, or at least as safe as BPG, for treating early syphilis. The investigators hypothesize that the recommended doxycycline regimen is not inferior to BPG and plan to test this hypothesis in a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients who, after the nature of the study has been explained to them, and before any protocol-specific procedures are performed, give informed consent in writing, in accordance with local regulatory requirements
* Patients with or without HIV infection and with syphilis infection in the early stages according to CDC criteria (primary syphilis, secondary syphilis and early latent syphilis of less than one year's duration)
* Patients with a positive non-treponemal assay result
* Patients available for participation and follow-up during the 6 months of the study
* Patients covered by the French health insurance system

Exclusion Criteria:

* Individuals with a history of known hypersensitivity to doxycycline or any other antibiotic of the tetracycline family, BPG (hypersensitivity to the active substance benzathine benzylpenicillin, to other penicillins, to soy phospholipids, peanuts or any of the excipients in the product ; history of severe immediate hypersensitivity reactions (eg anaphylaxis) to other beta-lactams (examples: cephalosporins, carbapenemes or monobactams), lidocaïne (hypersensitivity to lidocaine hydrochloride, amide-linked local anesthetics, or any of the excipients listed in SPC) and / or any of the excipients of the specialties used in the study
* Patients with a negative non-treponemal assay result
* Patients receiving an anticoagulant therapy
* Individuals with contraindications for either of the study drugs
* Individuals treated with retinoids by general route
* Individuals with early and late neurosyphilis
* Individuals requiring doxycycline treatment
* Individuals with late syphilis, whether or not latent (e.g. cutaneous)
* Individuals with thrombocytopenia or coagulation disorders contraindicating intramuscular injections
* Women who are pregnant or breast-feeding, or of childbearing age not using or planning to use acceptable birth control measures;
* Individuals under a measure of legal protection or unable to consent
* Individuals participating in any clinical trial with another investigational product in the 28 days preceding the first study visit or intending to participate in another clinical study at any time during the course of this study.
* Recent exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Demonstrate, with a high level of evidence, that doxycycline, administered orally at a dose of 100 mg bid for 14 days, is non-inferior to a single intramuscular injection of 2.4 million IU BPG for the treatment of early syphilis | 6 months
  Assessed on the basis of a four-fold decrease in titer in the non-treponemal assay (VDRL or RPR) at month 6 (commonly used to define cure in real-life settings) or a subsequent negative result in the non-treponemal test if the original test gave a results of 1/2 at inclusion.

SECONDARY OUTCOMES:
Evaluate tolerance to the two regimens in terms of severe adverse events (SAEs) | 6 months
  SAEs will be reported to the study sponsor
  * Photosentive reactions will be classified as minor, moderate, severe or very severe
  * Immediate hypersensitivity reaction will be classified as urticarial, angioedema or anaphylactic shock
  Jarisch-Herxeimer reactions will be evaluated at visit 1 (14 days ± 2 days)
Evaluate adherence to the doxycycline regimen | 6 months
  Adherence to doxycycline treatment will be evaluated on the basis of:
  * A tablet count at visit 1 (14 days ± 2 days)
  * The noting of tablet intake in the diary for the 14 days of the treatment period
Evaluate the impact of the two regimens on other STDs at month 6 | 6 months
  * PCR for CT, MG and NG will be performed systematically at month 6 on urine, or specimens from the throat or anus, depending on the sexual risk factors of the subject
  * HIV, hepatitis B serology, hepatitis C serology
demonstrate that doxycycline is non-inferior to a single intramuscular injection of BPG in titer in the non-treponemal assay (VDRL or RPR) | 3 months
  Response will be defined as a four-fold decrease (2 dilutions) in titer in the non-treponemal assay (VDRL or RPR) at month 6 relative to the assay performed before treatment. The two assays (before treatment and at month 6) should be performed in the same laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas DUPIN, PhD & MD, Principal Investigator — APHP Assistance Publique des Hôpitaux de Paris
Locations (7):
- France (7):
  - CHRU Jean Minjoz, Besançon
  - Hôpital Henri Mondor, Créteil
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Hotel Dieu, Paris
  - Hôpital Saint Louis - GeGIDD, Paris
  - Hôpital Saint Louis - SMIT, Paris
  - CHU Toulouse - Hôpital de la Grave - GeGIDD, Toulouse

IPD SHARING:
Plan to Share IPD: No